CLINICAL TRIAL: NCT07264426
Title: Real-World Efgartigimod Effectiveness in CIDP: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Other Study IDs: ARGX-113-NIS-2501
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy; CIDP; CIDP (Chronic Inflammatory Demyelinating Polyradiculoneuropathy)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — Efgartigimod treatment per country-specific label for the treatment of CIDP

SUMMARY:
The aims of this study are to assess the real-world effectiveness of efgartigimod in treating chronic inflammatory demyelinating polyradiculoneuropathy (CIDP), describe the "treatment journey" of participants with CIDP, and assess the utilization of health care services among adult participants with CIDP who initiate treatment with efgartigimod.

As this is a noninterventional study, treatment choices and decisions will be left to the discretion of participants and their physicians, according to the standard of care.

Each participant will be prospectively followed for up to 2 years from the date of initial administration of efgartigimod.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at time of providing informed consent
* Diagnosed with CIDP
* Planned to be receiving efgartigimod treatment within the CIDP treatment label of efgartigimod in the participant's respective country
* Efgartigimod treatment-naïve at time of screening

Exclusion Criteria:

* Polyradiculoneuropathy due to any other cause(s)
* Current participation in any interventional clinical study at time of screening, or planned participation before initiation of efgartigimod

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CIDP participants considered to be initiating efgartigimod treatment per country-specific label for the treatment of CIDP
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Change in aINCAT score over time | Up to 2 years and 3 months
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change in I-RODS score over time | Up to 2 years and 3 months
  Inflammatory Rasch-built Overall Disability Scale (I-RODS) assesses the limitations of activities and social participation in patients with inflammatory neuropathies like CIDP.
Change in grip strength over time | Up to 2 years and 3 months
Change in EQ-5D value from index date over time | Up to 2 years and 3 months
  The EQ-5D-5L questionnaire is a patient-reported outcome measure, ranging 0 to 100 (lower score, worse outcome)

CONTACTS AND LOCATIONS:
Locations (18):
- PPD Virtual, Wilmington, North Carolina, United States
- Germany (17):
  - Jüdisches Krankenhaus Berlin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Neurologie Neuer Wall - Dr.Bredow & Partner, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Gießen und Marburg GmbH - Standort Marburg, Marburg
  - Mühlenkreiskliniken - Johannes Wesling Klinikum Minden, Minden
  - Friedrich-Baur-Institute München, München
  - Immanuel Klinik Rüdersdorf, Rüdersdorf
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No